CLINICAL TRIAL: NCT01556061
Title: Comparison of Storz C-MAC and D-MAC Orotracheal Intubation Systems in Morbidly Obese Patients - A Prospective Randomized Crossover Trial
Brief Title: Comparison of Storz C-MAC and D-MAC Orotracheal Intubation Systems in Morbidly Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Davide Cattano, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-10-0573
Record Dates: First submitted 2012-03-01; First posted 2012-03-16 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-04

CONDITIONS: Obesity
Keywords: Laryngoscopy; Airway Management; Intubation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-MAC video laryngoscopy (Experimental): The Dblade is used to perfom laryngoscopy first but second laryngoscopy and intubation is performed with CMAC blade.
  Interventions: Device: DMAC; Device: CMAC
- C-MAC video laryngoscopy (Active Comparator): The CMAC blade is used to perfom laryngoscopy first but second laryngoscopy and intubation is performed with D-blade
  Interventions: Device: DMAC; Device: CMAC

INTERVENTIONS:
Device: DMAC — The D blade will constitute the experimental treatment and in a cross over fashion will be tested against CMAC blade
  Other Names: D-Blade CMAC system
Device: CMAC — The CMAC Blade will constitute the active comparator treatment and in a cross over fashion will be tested against D-blade
  Other Names: CMAC blade

SUMMARY:
The investigators hypothesize that the D-MAC (Dblade with C-MAC system) may be a suitable alternative device for difficult laryngoscopy and tracheal intubation in morbidly obese patients. The D-MAC will enable superior view of the glottic structures as well as easier endotracheal intubations than the C-MAC blade. This is the first study to investigate the individual and comparative performances of C-MAC and D-MAC in this patient cohort.

DETAILED DESCRIPTION:
Since the introduction of laryngoscopy, blades have undergone design innovations with the goal of improving laryngeal visualization and successful tracheal intubation because difficult intubation may be encountered even in patients with favorable anatomy.

Failed intubation shows occurrence in 0.05% of surgical patients and in 0.13% to 0.35% of obstetric and obese patients and the incidence of unsuspected difficult intubation is estimated to be higher at approximately 3%, with poor airway visualization being a major contributing factor.

Moreover airway management in the obese patient population requires special consideration. An increased BMI is associated with reduced posterior airway space and improper mask ventilation, both of which may lead to rapid development of hypoxemia and possible desaturation immediately after anesthetic induction.

As the prevalence of obesity has increased from 23% in 1992 to 33.8% in 2008 and an estimated 140,000 surgical bariatric cases are performed in the U.S., anesthesiologists face challenges of airway management in this population.

The main advantage of video intubation is provision of superior views compared to traditional laryngoscopy.

This study is designed to determine preliminarily the efficacy of the the D-BLADE [D-MAC] intubation systems compared to C-MAC in the bariatric population. The hypothesis is that D-MAC will enable superior view of the glottic structures as well as easier endotracheal intubations than the C-MAC blade.

A. General Study Design- The study will include a total of 50 morbidly obese patients (BMI ≥ 40kg/m2) scheduled for elective surgery (bariatric, gynecological, urological, general abdominal and otorhinolaryngology) at Memorial Hermann Hospital.

All patients will be intubated using conventional endotracheal tubes and preferably without any alternative aid to intubation. Patient will be followed for the time they will spend in the operating block (from the airway assessment time to the time of PACU discharge).

In the operating room, ASA standard monitoring devices will be applied: a pulse oximeter, a 3 lead ECG, and a blood pressure cuff (or invasive blood pressure depending on the patients' conditions). Pre-induction baseline measurements of blood pressure, heart rate, percent oxygen saturation and end tidal CO2 will be made. Patients will be positioned in a head elevated position (RAMP or TROOP pillow) and pre-oxygenated for 5 minutes. One set of pre-insertion vital signs (after induction) will be obtained. From the time anesthetic induction is begun until five minutes after the patient has been successfully intubated, five sets of vital signs will be recorded at one minute intervals. General anesthesia will be induced by bolus administration of propofol (2-3 mg/kg), fentanyl (2 mcg/kg), and succinylcholine (1mg/kg) per ideal body weight (assuming an ideal BMI of 32 kg/m2 up to a BMI of 50 kg/m2 and an ideal BMI 35 kg/m2 over 50 kg/m2. A rapid sequence induction (RSI) will be performed. RSI will be achieved with suxamethonium.The lungs will be mechanically ventilated with a semi-closed circle system to maintain an end-tidal CO2 near 35 mmHg. Patients' lungs will be ventilated via face-mask for 3 minutes with 100% oxygen until the patient is completely relaxed.

A ll investigators (residents and attending) will be trained based on manufacturer recommendations, and each resident will perform at least 3 intubations with the C-MAC and D-MAC video laryngoscope prior to enlisting any patients for the study. Intubations will be performed by 2nd and 3rd year (CA-2 and CA-3) residents. Size 3 blades of CMAC will be utilized in all cases (a size 4 will be available if necessary).

A computer-generated list will randomize the order of C-MAC and D-MAC to prevent bias. The resident will use either the C-MAC first followed by the D-MAC, or viceversa, and will declare the Cormack-Lehane Scale score for each method. Intubation will be attempted after the second laryngoscopy technique being used. External neck pressure may be applied by an assistant to improve laryngeal exposure. Any external manipulation will be recorded, and the optimal view obtained and the time required to obtain it for each method will be recorded.

The resident will have only one attempt each for C-MAC and D-MAC laryngoscopy. If the first attempt is unsuccessful, the attending anesthesiologist will take one more attempt for that particular method, C-MAC or D-MAC. The number of attempts (maximum 4 total as defined by reinsertion of either the blade or endotracheal tube), time required to obtain optimum view, CL score of view, and time required to intubate will all be recorded. Intubation time is defined by time from which the anesthesiologist has ETT in hand to when the ETT cuff passes distally through vocal cords. If unsuccessful, the direct laryngoscopy/flexible fiberoptic laryngoscopy will be performed to intubate the trachea. If more than 4 attempts are needed, or if the anesthesiologist discontinues use of the video laryngoscope, the case will be considered a failure. The resident's subjective opinion on laryngoscopy and intubation difficulty level (from 1 = Extremely Easy, to 5 = Extremely Difficult) will also be recorded.

In order to maintain patient safety all intubation attempts will be performed within the safety apnea time or time for oxygen blood saturation to drop to 92%.

B. Measurements Pre-operatively, morphometric characteristics of all patients will be recorded: Mallampati score, adequacy of neck mobility, neck circumference, thyromental distance, sternomental distance, and interincisor gap distance.

Degree of irritation: Following intubation in either group, the appearance of oropharynx, pharynx, epiglottis, and arytenoids will be checked. The presence of abrasions, bleeding, redness, perforation or other signs of tissue or dental injury will be recorded. Also, the patient's subjective report of soreness, hoarseness, or dysphagia post-operatively will be recorded as well.

DATA ANALYSIS:

This investigation will serve as preliminary study to determine if there is an improved rate of airway view during C-MAC or D-MAC video laryngoscopy. The study will have a time frame of 12 months. Data will be summarized using mean ± SD, median and interquantile, and frequency (%) for discrete variables by each group. Appropriate tests like t-test, ANOVA, chi-squared, and Fischer tests will be used to compare the mean primary outcome variable, duration of desaturation, between two groups after adjusting the effects of risk factors.

For the secondary outcome variables, appropriate tests like t-test, ANOVA, or the chi-squared tests will be performed to compare the continuous variables between two groups to compare the percentage of discrete outcome variables between two groups.

Statistical analyses will be conducted using STATA 10.0 College Station, TX and a p-value < 0.05 will be considered as statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* ASA I-III
* BMI ≥ 40 kg/m2

Exclusion Criteria:

* Necessary awake intubation
* Mallampati IV
* < 2 finger breath or 4 cm mouth opening
* Previous history of difficult intubation
* ASA IV-V
* Unstable cervical, thoracic and/or lumbar fracture
* Known history of congestive heart failure or a severe disease that alters pulmonary mechanics (e.g. chronic obstructive pulmonary disease, restrictive lung diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, MD, PhD, Principal Investigator — University Of Texas at Houston Medical School
Locations (1):
- Memorial Hermann Hospital-TMC, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dates of the recruitment period were 6/1/11 -12/12/11. Patients were recruited in the Preoperative Day Surgery area and preoperative Holding Unit.
Pre-assignment Details: No enrolled patients were excluded from the study.
Groups:
- C-MAC First, Then DMAC Video Laryngoscopy: C-MAC video laryngoscope (Intubation) : Patients assigned to this arm will have a first laryngoscopy with C-MAC video laryngoscope then a second laryngoscopy with the D-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with D-MAC laryngoscope.
- D-MAC First, Then CMAC Video Laryngoscopy: D-MAC video laryngoscope (Intubation) : Patients assigned to this arm will have a first laryngoscopy with D-MAC video laryngoscope then a second laryngoscopy with the C-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with C-MAC laryngoscope.
Period: Overall Study
Arm/Group | C-MAC First, Then DMAC Video Laryngoscopy | D-MAC First, Then CMAC Video Laryngoscopy
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- D-MAC First, Then C-MAC Video Laryngoscopy: D-MAC video laryngoscope (Intubation) : Patients assigned to this arm will have a first laryngoscopy with D-MAC video laryngoscope then a second laryngoscopy with the C-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with C-MAC laryngoscope.
- Total: Total of all reporting groups
Arm/Group | C-MAC First, Then DMAC Video Laryngoscopy | D-MAC First, Then C-MAC Video Laryngoscopy | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (11.0) | 46.2 (11.2) | 44.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time for Intubation
Description: Time taken for successful placement of endotracheal tube after a successful laryngoscopy. Typically a successful laryngoscopy will range from few seconds to no more than 90 seconds. A successful intubation will not range more than 90 seconds.
Time Frame: 90 seconds
Population: The unit of measure of time in seconds from D-MAC larynogoscopy to intubation in the (C-MAC Laryngoscopy First, Then DMAC Video Laryngoscopy) group and from C-MAC laryngoscopy to intubation in the (D-MAC Laryngoscopy First, Then C-MAC Video Laryngoscopy) group.
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- C-MAC Laryngoscopy First, Then DMAC Video Laryngoscopy: C-MAC video laryngoscope (D-MAC Intubation) : Patients assigned to this arm will have a first laryngoscopy with C-MAC video laryngoscope then a second laryngoscopy with the D-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with D-MAC laryngoscope.
- D-MAC Laryngoscopy First, Then C-MAC Video Laryngoscopy: D-MAC video laryngoscope (C-MAC Intubation) : Patients assigned to this arm will have a first laryngoscopy with D-MAC video laryngoscope then a second laryngoscopy with the C-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with C-MAC laryngoscope.
Arm/Group | C-MAC Laryngoscopy First, Then DMAC Video Laryngoscopy | D-MAC Laryngoscopy First, Then C-MAC Video Laryngoscopy
Number analyzed (Participants) | 25 | 25
seconds | 9 [5.85 to 13.95] | 7.3 [5.35 to 13.45]

2. Secondary Outcome: First Laryngoscopy
Description: Patients underwent laryngoscopy first with their assigned randomized laryngoscope. Time measured was from the time from the moment the anesthesiologist had the laryngoscope in hand to time to optimal visualization of vocal cords.
Time Frame: 30 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- C-MAC Video Laryngoscopy: C-MAC video laryngoscope (D-MAC Intubation) : Patients assigned to this arm will have a first laryngoscopy with C-MAC video laryngoscope then a second laryngoscopy with the D-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with D-MAC laryngoscope.
- D-MAC Video Laryngoscopy: D-MAC video laryngoscope (C-MAC Intubation) : Patients assigned to this arm will have a first laryngoscopy with D-MAC video laryngoscope then a second laryngoscopy with the C-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with C-MAC laryngoscope.
Arm/Group | C-MAC Video Laryngoscopy | D-MAC Video Laryngoscopy
Number analyzed (Participants) | 25 | 25
seconds | 6.7 [4.45 to 9.7] | 7.2 [4.82 to 9.95]

3. Secondary Outcome: Second Laryngoscopy
Description: A second laryngoscopy will be performed in patients with the video laryngoscope from the other group. Patients will be intubated after second laryngoscopy with with this same video laryngoscope.
Time Frame: 30 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | C-MAC Video Laryngoscopy | D-MAC Video Laryngoscopy
Number analyzed (Participants) | 25 | 25
seconds | 6.7 [4.2 to 9.1] | 5.5 [4.04 to 9.4]

ADVERSE EVENTS:
Groups:
- DMAC Laryngoscopy First, Then C-MAC Video Laryngoscopy: D-MAC video laryngoscope (C-MAC Intubation) : Patients assigned to this arm will have a first laryngoscopy with D-MAC video laryngoscope then a second laryngoscopy with the C-MAC video laryngoscope. Patients will be intubated after second laryngoscopy with C-MAC laryngoscope.
Arm/Group | C-MAC Laryngoscopy First, Then DMAC Video Laryngoscopy | DMAC Laryngoscopy First, Then C-MAC Video Laryngoscopy
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No